CLINICAL TRIAL: NCT04013568
Title: A Pilot Study: The Effect of Longitudinal Exercise Programming in Breast Cancer Patients
Brief Title: Exercise Post-Diagnosis of Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Rehabilitation Hospital of the Pacific (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fukui-2019-1
Record Dates: First submitted 2019-06-14; First posted 2019-07-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants choose the initial intervention (12-week exercise program (Group1) vs monitoring (Group2)).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Agree to Exercise Program (Active Comparator): 12-week exercise program
  Interventions: Other: Exercise
- Group 2 - Declines Exercise Program (No Intervention): Same biometric and biomarker assessment at as Group 1 (at baseline, after 12 weeks and annually) however they will not participate in the exercise sessions

INTERVENTIONS:
Other: Exercise — First Intervention 12-week exercise program, 3 days/week, 90min exercise sessions at the Rehabilitation Hospital of the Pacific. Private or semi-private (1:1 or 2:1 ratio participant to instructor) sessions, led by Kinesiology students
  Second Intervention- 12-week exercise program, 2 days/week, 90min exercise sessions at the Rehabilitation Hospital of the Pacific. Group Fitness Classes
  Arms: Group 1 - Agree to Exercise Program

SUMMARY:
The investigators are doing this study to determine if there are body composition changes after a 12-week exercise program in breast cancer patients and determine what factors contribute to sustained physical activity after the 12-week exercise program intervention.

DETAILED DESCRIPTION:
The study is enrolling breast cancer patients up to 2 years after their diagnosis in a 12-week exercise program. The participants will either participate in: Group 1-participating in an exercise program with biometric evaluations or Group 2-biometric evaluations but not participating in the exercise program. At the end of the 12-week exercise program, participants in Group 1 will be randomized to either: a) continuing with exercise group classes or b) continuing with exercise individual classes. Both Group 1a and 1b participants will be followed for the remainder of the year and be evaluated for continued physical activity. All Group study participants' biometrics will be assessed at baseline and at the end of 12-weeks, with continued annual medical review follow-up for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of breast cancer (within the past 2 years, any subtype, stage I-III)
* Can be undergoing neo/adjuvant treatment (surgery, chemotherapy, radiation or endocrine therapy)
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing scheduled exercise sessions, completing questionnaires and biometric/biomarker studies
* Participant must be able to lie flat on their back for up to 10 minutes
* Participant must be able to stand without aid for at least 2 minutes

Exclusion Criteria:

* Participant with breast cancer recurrence
* Metastatic breast cancer
* Uncontrolled psychiatric disorder that can affect self-assessment
* Pregnant patient
* Participants with any internal artifact (e.g. pacemakers, internal fixation, arthroplasty) or other physical impairment that would alter the body composition assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Fat mass | 1 day
  Measure fat mass (arms, legs, trunk and total) in kg using Dual energy X-ray absorptiometry (DXA) data
Isometric peak torque | 1 day
  Measure the peak torque value generated during isometric knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device
Lean mass | 1 day
  Measure lean mass (arms, legs, trunk and total) in kg using Dual energy X-ray absorptiometry (DXA) data
Bone mass | 1 day
  Measure bone mass (arms, legs, trunk and total) in kg using Dual energy X-ray absorptiometry (DXA) data
Waist to Hip ratio (WHR) from manual tape measurement | 1 day
  Manual physical anthropometry of waist and hip circumferences
Automatic 3D optical (3DO) scan measurement: girth measurement | 1 day
  Automated 3DO measurements generate the following: girth in cm measurements across the whole body
Muscle Function | 1 day
  Measure the peak torque value generated during isometric knee extension/flexion movement evaluation at 60 degrees will be assessed with the HUMAC NORM device
Percent fat | 1 day
  Percent fat (arms, legs, trunk and total) using Dual energy X-ray absorptiometry (DXA) data
Automatic 3D optical (3DO) scan measurement: length measurement | 1 day
  Automated 3DO measurements generate the following: length in cm measurements across the whole body
Automatic 3D optical (3DO) scan measurement: volume measurement | 1 day
  Automated 3DO measurements generate the following: volume in cm measurements across the whole body
Bone Mineral Density (spine and total) using Dual energy X-ray absorptiometry (DXA) data | 1 day
  Bone Mineral Density (spine and total) using Dual energy X-ray absorptiometry (DXA) data

SECONDARY OUTCOMES:
Recurrence Free Survival | 5 years
  obtained from last physician note
BIBCQ-Body Image After Breast Cancer questionnaire | 5 years
  45 items
BFI-Brief Fatigue Innovatory questionnaire | 5 years
  9 items
PHQ-9- Patient Health (Depression) questionnaire | 5 years
  9 items
FACT-G-Functional Assessment of Cancer Therapy-General (Comorbidities)questionnaire | 5 years
  27 items
Diet History Questionnaire II | 5 years
  Self-reported energy intake, measured as kcal/day
Biomarkers | 5 years
  Adipokines: leptin, HMW-high molecular weight adiponectin, PAI1-plasminogen activator inhibitor
  Cytokines & Inflammation: TNF-tumor necrosis factor α, IL-interleukin 1β, IL2, IL4, IL5, IL6, IL8, IL10, interferon, CRP-C reactive protein, uric acid, cortisol
  Insulin Resistance & IGFs: glucose, insulin, Hb-hemoglobin A1C, IGF-insulin growth factor 1, IGFBP-insulin like growth factor binding protein 1-3
  Sex Steroid Hormones: total estradiol & estrone, total testosterone, SHBG-sex hormone-binding globulin (for free estradiol and free testosterone will be derived)
  Lipid Profile & Lipid-soluble Micronutrients: TG-triglycerides , total cholesterol, HDLC-high density lipoprotein cholesterol , free fatty acids, lycopene, 25OH-vitamin D3, alpha-tocopherol
  Liver Enzymes: ALT-alanine aminotransferase
  Neuropeptides & Gut Hormones: ghrelin
  MOTS-mitochondrial derived peptide-c

CONTACTS AND LOCATIONS:
Overall Officials: Jami Fukui, MD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No